CLINICAL TRIAL: NCT02137499
Title: Venous Insufficiency and Neuromuscular Stimulation
Acronym: VeINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/WM/0027; CR02072 (Other: Imperial College London)
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Chronic Venous Disease; Venous Insufficiency; Deep Venous Obstruction
Keywords: Deep venous obstruction; Venous insufficiency
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy subjects (Active Comparator): Healthy subjects, free from vascular disease
  Interventions: Device: geko device
- Superficial venous insufficiency (Experimental): Clinically symptomatic and ultrasound evidence of superficial venous insufficiency
  Interventions: Device: geko device
- Deep venous insufficiency (Experimental): Clinically symptomatic and ultrasound evidence of deep venous insufficiency
  Interventions: Device: geko device
- Deep venous obstruction (Experimental): Clinically symptomatic and ultrasound evidence of deep venous obstruction
  Interventions: Device: geko device

INTERVENTIONS:
Device: geko device — Small transcutaneous electrical stimulator. Manufactured in UK by Firstkind UK Ltd, and licensed for use in humans

SUMMARY:
The investigators will be evaluating the immediate and longer term effect of treatment with a medical device on the symptoms of chronic venous disease.

DETAILED DESCRIPTION:
STUDY AIMS

1. To obtain ultrasound blood flow and velocity measurements in the leg to compare the hemodynamic profiles obtained using a neuromuscular stimulation device with those obtained at rest.
2. To ascertain if a 6 week protocol of electrical neurostimulation of the muscle pumps in the leg and foot can reduce clinical symptoms and improve quality of life.

METHODS Controlled interventional trial. Group 1 (10 subjects) will be healthy subjects with no clinical venous disease. Subjects with venous incompetence to be recruited into one of three groups. Group 2 (10 subjects) will have superficial venous incompetence; Group 3 (10 subjects) will have deep venous incompetence; Group 4 (10 subjects) will have deep vein occlusion. These will be clinical diagnoses confirmed with duplex ultrasound.

The device used in this study will be the geko™ T-1 device (Firstkind Ltd, UK). A geko™ device will be fitted to each leg. The device stimulation level is set to the minimum level that can achieve the desired response (outward and upward twitching of the foot when raised from the ground).

ENDPOINTS Primary end-point

* Increase in venous flow Secondary end points
* Improvement in clinical symptoms at 6 weeks, as judged by questionnaire
* Reduction in absolute leg diameter and volume at 6 weeks

ELIGIBILITY:
Group 1

* Inclusion criteria - 18+ years old, 17<BMI<30
* Exclusion criteria - Heart/lung/kidney failure, pregnancy, diagnosis of peripheral vascular disease, previous VTE, ABPI<0.9, active infection, previous leg fracture or metal implant in leg

Group 2

* Inclusion criteria - 18+ years old, 17<BMI<30, clinical diagnosis of superficial venous insufficiency (CEAP C2-6) confirmed with duplex US
* Exclusion criteria - Heart/lung/kidney failure, pregnancy, ABPI<0.9, active infection, previous leg fracture or metal implant in leg

Group 3

* Inclusion criteria - 18+ years old, 17<BMI<30, clinical diagnosis of deep venous insufficiency (CEAP C2-6) confirmed with duplex US
* Exclusion criteria - Heart/lung/kidney failure, pregnancy, ABPI<0.9, active infection, previous leg fracture or metal implant in leg

Group 4

* Inclusion criteria - 18+ years old, 17<BMI<30, clinical diagnosis of deep venous obstruction confirmed with duplex US
* Exclusion criteria - Heart/lung/kidney failure, pregnancy, ABPI<0.9, active infection, previous leg fracture or metal implant in leg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alun Davies, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, Hammersmith, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams KJ, Moore HM, Ellis M, Davies AH. Pilot Trial of Neuromuscular Stimulation in Human Subjects with Chronic Venous Disease. Vasc Health Risk Manag. 2021 Dec 1;17:771-778. doi: 10.2147/VHRM.S320883. eCollection 2021. PMID 34880620

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Subjects: Healthy participants treated with Small transcutaneous electrical stimulator
- Superficial Venous Insufficiency: Participants with Superficial venous insufficiency treated with Small transcutaneous electrical stimulator
- Deep Venous Insufficiency: Participant with Deep venous insufficiency treated with Small transcutaneous electrical stimulator
- Deep Venous Obstruction: Participant with Deep venous obstruction treated with Small transcutaneous electrical stimulator
Period: Overall Study
Arm/Group | Healthy Subjects | Superficial Venous Insufficiency | Deep Venous Insufficiency | Deep Venous Obstruction
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Deep Venous Insufficiency: Participants with Deep venous insufficiency treated with Small transcutaneous electrical stimulator
- Deep Venous Obstruction: Participants with Deep venous obstruction treated with Small transcutaneous electrical stimulator
- Total: Total of all reporting groups
Arm/Group | Healthy Subjects | Superficial Venous Insufficiency | Deep Venous Insufficiency | Deep Venous Obstruction | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (10) | 55 (15) | 58.6 (18) | 53.2 (16) | 56 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 2 | 3 | 16
  Male | 5 | 4 | 8 | 7 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change of Haemodynamic Flow
Description: Doppler ultrasound measurements of femoral venous blood flow. The volume flow rate in blood vessel can be calculated by multiplying the cross-sectional area of the blood vessel by the mean velocity of the blood within it.
Time Frame: baseline, 20 minutes
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Healthy Subjects | Superficial Venous Insufficiency | Deep Venous Insufficiency | Deep Venous Obstruction
Number analyzed (Participants) | 10 | 10 | 10 | 10
% change
  Peak velocity | 34.8 [-4 to 81] | 62.8 [25 to 138] | 9 [-10 to 84] | 14.8 [-8 to 51]
  TAMV time-averaged mean velocity | -14.2 [-30 to 55] | 28.1 [-2 to 111] | 28.2 [-30 to 66] | -5.1 [-28 to 35]
  Volume flow | -22.5 [-40 to 40] | 37.5 [-10 to 172] | 17.4 [1 to 49] | 5.9 [-11 to 21]

2. Secondary Outcome: Improvement in Venous Symptoms
Description: Clinical symptoms will be measured using questionnaires (AVVQ, VCSS)
Time Frame: 6 weeks
Population: Data not collected
Arm/Group | Healthy Subjects | Superficial Venous Insufficiency | Deep Venous Insufficiency | Deep Venous Obstruction
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Leg Volume
Description: Measured using ankle and calf circumference, and multiplying using "inverted cone" method
Time Frame: 6 weeks
Population: Data not collected
Arm/Group | Healthy Subjects | Superficial Venous Insufficiency | Deep Venous Insufficiency | Deep Venous Obstruction
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Healthy Subjects | Superficial Venous Insufficiency | Deep Venous Insufficiency | Deep Venous Obstruction
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes